CLINICAL TRIAL: NCT05712629
Title: The Effect of Functional Bread Dadih During Pregnancy and Health Outcomes
Brief Title: The Effect of Functional Bread Dadih on Microbiota Profile of Weight Increase Pregnant Women and Infant Birth Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andalas University (Other)
Collaborators: National Institute of Health Research and Development, Ministry of Health Republic of Indonesia (Other)
Responsible Party: Principal Investigator, Dr. Helmizar, SKM, M.Biomed, Dr. Helmizar, SKM, M.Biomed, Andalas University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HL
Record Dates: First submitted 2023-01-03; First posted 2023-02-03 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Birth Weight; Pregnancy Weight Gain
Keywords: Functional Bread; Weight Increase; Infant Weight
MeSH Terms: conditions — Birth Weight; Gestational Weight Gain; Weight Gain | interventions — Bread

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Responden Intervention (Active Comparator): Arm 1 (Interventional) : Respondent has given bread with composit flour and vla with dadiah. pregnant women received 1 pieces bread containing 50 gram provide total fat 4 gram, protein 5 gram, carbohydrate 23.8 gram, Fe 2 mg, 2150 kcal and vla dadiah containing 30 gram provide 308 kcal.
  Interventions: Other: Bread and vla dadiah
- Responden Placebo (Placebo Comparator): Arm 2 (Placebo) : Respondent has given bread with original flour (wheat flour) and vla original without dadiah. pregnant women received 1 pieces bread containing 50 gram and vla containing 30 gram.
  Interventions: Other: Bread and vla without dadiah

INTERVENTIONS:
Other: Bread and vla dadiah — Consumption bread and vla dadiah to pregnant women 1 Pieces a day during 12 weeks.
  Arms: Responden Intervention
Other: Bread and vla without dadiah — Consumption bread and vla without dadiah to pregnant women 1 Pieces a day during 12 weeks.
  Arms: Responden Placebo

SUMMARY:
The aims of study to determine the effect of giving functional bread and dadih's vla on weight gain of pregnant women and birth weight of babies.

DETAILED DESCRIPTION:
Dadih contains BAL 108 CFU/ml which is probiotic. Consumption of functional bread and dadih's vla during pregnancy can improve the composition of the gut microbiota so that it can increase maternal weight and provide adequate nutrition during pregnancy. Good nutrient absorption can support good nutritional status and weight in babies who are born. This study aims to determine the effect of giving functional bread and dadih's vla on weight gain of pregnant women and birth weight of babies.

This study used a randomized controlled trial (RCT) design with a population of all pregnant women in the Kuranji, Nanggalo and Andalas Health Centers. The sample consisted of 88 people and was divided into two groups, namely the intervention group and the control group. Each amounted to 44 samples. The sample selection used the double-blind method and randomized controlled trial (RCT) research design. The intervention started at about 12-20 weeks of gestation and continued until just before the time of delivery. In the third trimester, subjects received healthy food, breastfeeding practices, and child development education to support mothers in maintaining their nutritional status, preparing exclusive breastfeeding, and optimizing child development.

Healthy babies born to mothers will be the focus of this study and followed up until the age of three months to assess their growth. The information includes the baby's health history after birth, anthropometric measurements, nutritional intake, and breastfeeding practices which are measured repeatedly in the first, second, and third months.

Data quality assurance is carried out through training starting from the period of data collection and supervision during and after data collection, including the data analysis process. This included training for enumerators, subjects and using a validated questionnaire for a group of subjects representing similar characteristics for this study. Data input and cleaning process will use excel and SPSS while for food intake data using NutriSurvey 2007. Data entry will be carried out by data collection officers after data collection. The data cleaning process includes removing outliers and regrouping multiple results that have similar meanings. The data will be interpreted as mean ± standard deviation if the data is normally distributed and the median (min-max) if the data is not normally distributed. Statistical analysis using SPSS 25 and data will be analyzed using univariate and bivariate analysis. Univariate analysis is used to describe characteristics and socio-demographics, medical history, pregnancy, and obstetric profiles of pregnant women. Numerical variables between groups will be analyzed using an Independent sample t-test if the data has normal distribution or the Mann Whitney test if the data distribution is not normal. Categorical variables between groups will be analyzed using Chi-square or Fisher test. Differences between birth and 3 months old follow up will be analyzed using independent t-tests if the data distribution has normal distribution or Mann Whitney test if the data distribution is not normal.

ELIGIBILITY:
Inclusion Criteria:

* Mothers with gestational 12 - 20 weeks
* Health Conditions
* Not moving home until delivery labour
* Not suffering from syndrome metabolic diseases

Exclusion Criteria:

* Not willing and signing an informed consent, and not willing to consume fungtional bread and dadih's vla or dadih sauce until delivery.
* Abortus

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Body Weight Pregnant Woman Measurement | 12 weeks
  Measuring Body Weight Pregnant Woman Baseline, 1St Measurement, 2nd Measurement, and 3rd Measurement (Weight in Kilograms)
Body Height Pregnant Woman Measurement | 12 weeks
  Measuring Body Height Pregnant Woman Baseline, 1St Measurement, 2nd Measurement, and 3rd Measurement (Height in Meters or Centimeters)
Body Mass Index Pregnant Woman Measurement | 12 weeks
  Measuring Body Height Pregnant Woman Baseline, 1St Measurement, 2nd Measurement, and 3rd Measurement (BMI in Kg/m^2)
Birth Weight of Infant Measurement | 9 months
  Measuring weight of infant (Weight in Grams)
Birth Length of Infant Measurement | 9 months
  Measuring Birth Length of infant (Length or height in Centimeters)

SECONDARY OUTCOMES:
Characteristic of Woman Pregnancy | 4 weeks
  Description of Characteristic respondent are Mother's tribe, mother's education, mother's job, mother's knowledge, family income, age, and gestational weeks

CONTACTS AND LOCATIONS:
Overall Officials: Helmizar Helmizar, DR, Principal Investigator — Nutrition Department Faculty of Universitas Andalas; Azrimaidaliza Azrimaidaliza, DR, Study Director — Department Nutrition Faculty of Universitas Andalas; Ferdinal Ferry, DR, Study Director — Department Obstetry and Gynecology of Universitas Andalas; Frima Elda, DR, Study Director — Department Nutrition Faculty of Universitas Andalas; Asrawati Asrawati, DR, Study Director — Department Pediatric of Universitas Andalas
Locations (1):
- Universitas Andalas, Padang, West Sumatera, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wijayanti, IA, Purwadi, P., & Thohari, I. (2017). The Effect of Adding Sago Flour to Yoghurt on the Physical Properties of Yoghurt Ice Cream. Journal of Animal Products Science and Technology (JITEK), 11(1), 38-45.
- [Background] Wijayanti, MDS, Thohari, I., & Purwadi, P. 2017. Quality of curd in goat's milk incubated on various kinds of bamboo. Journal of Animal Products Science and Technology (JITEK), 11(1), 22-37.
- [Result] Astuti, S.D., Andarwulan, N., Hariyadi, P. and Agustia, F.C., 2014. Formulasi dan karakterisasi cake berbasis tepung komposit organik kacang merah, kedelai, dan jagung. Jurnal Aplikasi Teknologi Pangan, 3(2).
- [Result] Black, R.E. and Hopkins Bloomberg, J., 2008. The lancet series on maternal and child Undernutrition, executive summary. Lancet, 371, pp.1-10.
- [Result] Brown KH, Peerson JM, Rivera J, Allen LH. Effect of supplemental zinc on the growth and serum zinc concentrations of prepubertal children: a meta-analysis of randomized controlled trials. Am J Clin Nutr. 2002 Jun;75(6):1062-71. doi: 10.1093/ajcn/75.6.1062. PMID 12036814
- [Result] Collado MC, Surono IS, Meriluoto J, Salminen S. Potential probiotic characteristics of Lactobacillus and Enterococcus strains isolated from traditional dadih fermented milk against pathogen intestinal colonization. J Food Prot. 2007 Mar;70(3):700-5. doi: 10.4315/0362-028x-70.3.700. PMID 17388062
- [Result] Caulfield, L.E., Huffman, S.L. and Piwoz, E.G., 1999. Interventions to improve intake of complementary foods by infants 6 to 12 months of age in developing countries: impact on growth and on the prevalence of malnutrition and potential contribution to child survival. Food and nutrition bulletin, 20(2), pp.183-200.
- [Result] Young Child Nutrition Working Group: Formulation Subgroup. Formulations for fortified complementary foods and supplements: review of successful products for improving the nutritional status of infants and young children. Food Nutr Bull. 2009 Jun;30(2 Suppl):S239-55. No abstract available. PMID 20496618
- [Result] Dijkhuizen MA, Wieringa FT, West CE, Martuti S, Muhilal. Effects of iron and zinc supplementation in Indonesian infants on micronutrient status and growth. J Nutr. 2001 Nov;131(11):2860-5. doi: 10.1093/jn/131.11.2860. PMID 11694609
- [Result] Fahmida U, Rumawas JS, Utomo B, Patmonodewo S, Schultink W. Zinc-iron, but not zinc-alone supplementation, increased linear growth of stunted infants with low haemoglobin. Asia Pac J Clin Nutr. 2007;16(2):301-9. PMID 17468087
- [Result] Helmizar H, Jalal F, Lipoeto NI, Achadi EL. Local food supplementation and psychosocial stimulation improve linear growth and cognitive development among Indonesian infants aged 6 to 9 months. Asia Pac J Clin Nutr. 2017 Jan;26(1):97-103. doi: 10.6133/apjcn.102015.10. PMID 28049268
- [Result] Hess SY, Lonnerdal B, Hotz C, Rivera JA, Brown KH. Recent advances in knowledge of zinc nutrition and human health. Food Nutr Bull. 2009 Mar;30(1 Suppl):S5-11. doi: 10.1177/15648265090301S102. PMID 19472599
- [Result] Hoj S, Fredholm M, Larsen NJ, Nielsen VH. Growth hormone gene polymorphism associated with selection for milk fat production in lines of cattle. Anim Genet. 1993 Apr;24(2):91-5. doi: 10.1111/j.1365-2052.1993.tb00246.x. PMID 7687103
- [Result] Khotimah, K. and Kusnadi, J., 2014. Antibacterial Activity of Probiotic Dates (Phoenix dactilyfera L.) Using Lacbobacillus plantarum and Lacbobacillus casei. J. Pangan Agroind, 2(3), pp.110-120.
- [Result] Efendi F, Chen CM, Kurniati A, Berliana SM. Determinants of utilization of antenatal care services among adolescent girls and young women in Indonesia. Women Health. 2017 May-Jun;57(5):614-629. doi: 10.1080/03630242.2016.1181136. Epub 2016 May 26. PMID 27230132
- [Result] Lozupone CA, Stombaugh JI, Gordon JI, Jansson JK, Knight R. Diversity, stability and resilience of the human gut microbiota. Nature. 2012 Sep 13;489(7415):220-30. doi: 10.1038/nature11550. PMID 22972295
- [Result] Ojofeitimi, E.O., Ogunjuyigbe, P.O., Sanusi, R.A., Orji, E.O., Akinlo, A., Liasu, S.A. and Owolabi, O.O., 2008. Poor dietary intake of energy and retinol among pregnant women: implications for pregnancy outcome in Southwest Nigeria. Pak. J. Nutr, 7(3), pp.480-484.
- [Result] Arnold, M., Rajagukguk, Y.V. and Gramza-Michałowska, A., 2021. Characterization of Dadih: Traditional Fermented Buffalo Milk of Minangkabau. Beverages, 7(3), p.60.
- [Result] Unayah, A., Estuti, W., Kunaepah, U., Studies, N., Tasikmalaya, P.K. and Barat, J., 2020. Use of Local Food Ingredients MOCAF (Modified Cassava Flour) and Rebon Planktonic Shrimp) in Cookies as an Alternative Supplementary Food for Children. International Journal of Innovation, Creativity and Change, pp.1035-1050.
- [Result] Surono IS. Traditional Indonesian dairy foods. Asia Pac J Clin Nutr. 2015;24 Suppl 1:S26-30. doi: 10.6133/apjcn.2015.24.s1.05. PMID 26715081
- [Result] Surono IS, Martono PD, Kameo S, Suradji EW, Koyama H. Effect of probiotic L. plantarum IS-10506 and zinc supplementation on humoral immune response and zinc status of Indonesian pre-school children. J Trace Elem Med Biol. 2014 Oct;28(4):465-9. doi: 10.1016/j.jtemb.2014.07.009. Epub 2014 Aug 2. PMID 25183688
- [Result] Shah, N.P., 2006. Health benefits of yogurt and fermented milks. Manufacturing yogurt and fermented milks, 327.
- [Result] UNICEF. Division of Communication and UNICEF., 2009. Tracking progress on child and maternal nutrition: a survival and development priority. Unicef.
- [Result] Yarandi SS, Peterson DA, Treisman GJ, Moran TH, Pasricha PJ. Modulatory Effects of Gut Microbiota on the Central Nervous System: How Gut Could Play a Role in Neuropsychiatric Health and Diseases. J Neurogastroenterol Motil. 2016 Apr 30;22(2):201-12. doi: 10.5056/jnm15146. PMID 27032544
- See also: Zinc-iron, but not zinc-alone supplementation, increased linear growth of stunted infants with low haemoglobin. Asia Pacific Journal of Clinical Nutrition, 16(2), pp.301-309. — https://citeseerx.ist.psu.edu/document?repid=rep1&type=pdf&doi=9bfddcc516734cbaa5b55d235971a1b213e146a8
- See also: Antibacterial Activity of Probiotic Dates (Phoenix dactilyfera L.) Using Lacbobacillus plantarum and Lacbobacillus casei. J. Pangan Agroind, 2(3), pp.110-120. — https://pdfs.semanticscholar.org/7934/f3e473c8024109718faafa08c70569ed06e2.pdf
- See also: Diversity, stability and resilience of the human gut microbiota. Nature, 489(7415), pp.220-230. — https://www.nature.com/articles/nature11550
- See also: Use of Local Food Ingredients MOCAF (Modified Cassava Flour) and Rebon Planktonic Shrimp) in Cookies as an Alternative Supplementary Food for Children. International — https://www.ijicc.net/images/vol_13/Iss_2/SC40_Unayah_2020_E_R.pdf
- See also: Effect of probiotic L. plantarum IS-10506 and zinc supplementation on humoral immune response and zinc status of Indonesian pre-school children. Journal of Trace Elements in Medic — https://pubmed.ncbi.nlm.nih.gov/25183688/
- See also: Tracking progress on child and maternal nutrition: a survival and development priority. Unicef. — https://books.google.com/books?hl=en&lr=&id=-qS8H55N7AUC&oi=fnd&pg=PA3&dq=UNICEF.+(2009).+Tracking+Progress+on+Child+and+Maternal+Nutrition:+A+survival+and+development+priority.+Unicef,+New+York.&ots=3e7Y6efUI1&sig=C2fqxBO5duWxQTVgWQPZdYGmvS8
- See also: Modulatory effects of gut microbiota on the central nervous system: how gut could play a role in neuropsychiatric health and diseases. Journal of neurogastroenterology an — https://pubmed.ncbi.nlm.nih.gov/27032544/

DOCUMENTS (1):
  • Study Protocol (2022-12-13): https://cdn.clinicaltrials.gov/large-docs/29/NCT05712629/Prot_000.pdf